CLINICAL TRIAL: NCT00891774
Title: An Open-label, Multi-Center, Prospective, Post Market Study to Assess the Safety and Effectiveness of EVOLENCE® in Facial Augmentation of Subjects With Fitzpatrick Skin Color Types IV, V, and VI
Brief Title: Post Market Safety Study and Effectiveness With Evolence in Subjects With Skin Color Types IV-VI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DP101 US-04; NCT00871988 (obsolete NCT alias)
Record Dates: First submitted 2009-04-30; First posted 2009-05-01 (Estimated); Results first posted 2011-05-13 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-01

CONDITIONS: Non Therapeutic Body Modification

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Device (Experimental): Treatment with EVOLENCE®
  Interventions: Device: EVOLENCE®

INTERVENTIONS:
Device: EVOLENCE® — Single injection of material into the mid-dermis of the wrinkle - Second 'touch-up' injection is permitted approximately 14-Days later if needed to achieve satisfactory results
  Other Names: Facial augmentation

SUMMARY:
Approximately 165 subjects with Fitzpatrick Skin Color Types IV, V, and VI and a moderate to deep wrinkle between the corner of the nose and the corner of the mouth, will be treated with EVOLENCE® (an approved collagen filler) to smooth and flatten that wrinkle. They will be observed for 6 months to establish safety of the product as it relates to scarring and changes in skin pigment, and long term effectiveness.

DETAILED DESCRIPTION:
This is an open-label, multi-center, prospective, postmarket study to assess the safety and effectiveness of EVOLENCE® (DP101) in Subjects with Fitzpatrick Skin Color Types IV, V, and VI seeking correction of bilateral facial wrinkles and folds of the nasolabial area.

The study will enroll and treat a total of 165 subjects with Fitzpatrick Skin Color Types IV, V and VI who have clinical evidence of moderate to deep bilateral wrinkles in the nasolabial area.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* moderate to deep wrinkle in the Naso-Labial fold
* Fitzpatrick Skin Type IV, V or VI

Exclusion Criteria:

* Pregnant or nursing females
* Hx of allergies to related products
* history of keloids, active skin disease, or previous augmentation of the treatment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2008-12-31 (Actual); Primary Completion 2009-11-30 (Actual); Study Completion 2009-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Shoshani, MD, Study Director — Colbar/OrthoDermatologics
Locations (11):
- United States (11):
  - The Vitiligo and Pigmentation Institute of Southern California, Los Angeles, California
  - Desert Dermatology Medical Associates, Rancho Mirage, California
  - Center for Dermatology and Dermatologic Surgery, Washington D.C., District of Columbia
  - Atlanta Dermatology Vein & Research Center, Alpharetta, Georgia
  - Denova Research, Chicago, Illinois
  - DuPage Medical Group Clinical Research, Naperville, Illinois
  - Callender Center for Clinical Research, Mitchellville, Maryland
  - The Boyd Gillard Institute of Aesthetic & Dermatology Surgery, Ypsilanti, Michigan
  - Image Dermatology, Montclair, New Jersey
  - Susan Taylor, Philadelphia, Pennsylvania
  - Tennessee Clinical Research, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Device
Started | 172
Completed | 158
Not Completed | 14
Not completed — Lost to Follow-up | 5
Not completed — Illness (Self/Mother) | 3
Not completed — Withdrawal by Subject | 2
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Arm/Group | Device
Number analyzed (Participants) | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 150
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18
  Not Hispanic or Latino | 154
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 135
  White | 17
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Count of Participants; unit: Participants]
  North America: United States | 172
Fitzpatrick Skin Tone [Count of Participants; unit: Participants]
  IV (Light Brown) | 54
  V (Brown) | 66
  VI (Dark Brown/Black) | 52

OUTCOME MEASURES:

1. Primary Outcome: Safety Endpoint
Description: Safety Endpoint includes three categories: 1) composite determination of success (no pigmentation change or keloid formation); 2) pigmentation changes; and 3) keloid formation
Time Frame: 6 months post injection
Measure: Number; unit: Participants
Arm/Group | Device
Number analyzed (Participants) | 172
Participants
  Success | 155
  Keloid Formation | 0
  Pigmentation Change | 3

2. Secondary Outcome: Reduction in Wrinkle Severity Score
Time Frame: Baseline, 1, 3 and 6 months post injection
Population: Sponsor made business decision to discontinue marketing of product in US and program was terminated before full analysis of results. No analysis was performed on Secondary Outcome Measures. Sincere efforts were made to obtain secondary outcome measure data; there is no longer access to these data and therefore no data can be reported.
Arm/Group | Device
Number analyzed (Participants) | 0

3. Secondary Outcome: Investigator's Satisfaction of the Overall Treatment
Time Frame: 1, 3 and 6 months post injection
Population: as for outcome 2
Arm/Group | Device
Number analyzed (Participants) | 0

4. Secondary Outcome: Subject's Satisfaction of the Overall Treatment
Time Frame: 1, 3 and 6 months post injection
Population: as for outcome 2
Arm/Group | Device
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Device
Serious Adverse Events (participants affected / at risk) | 3/158
Other Adverse Events (participants affected / at risk) | 154/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Device (N=158)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Enlarging Multifibroid Uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder Failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Device (N=154)
Administration Site Conditions (General disorders) | 154
Oral or Upper Respiratory Infections (Infections and infestations) | 12
Erythema (Skin and subcutaneous tissue disorders) | 17
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 12

LIMITATIONS AND CAVEATS:
Sponsor discontinued US marketing of product; program terminated. No analysis performed on Secondary Measures. Sincere efforts were made to obtain secondary measure data; there is no longer access to these data and therefore no data can be reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No paper that incorporates Sponsor Confidential Information will be submitted for publication without Sponsor's prior written consent. The Institution will provide Sponsor with at least sixty (60) days for review of a manuscript, and if requested in writing, the Institution and Principal Investigators will withhold such publication for up to an additional sixty (60) days to allow for filing of a patent application.